CLINICAL TRIAL: NCT00904228
Title: Effectiveness of Plastic Lined Hats for Prevention of Hypothermia in Premature Newborns in the Delivery Room
Brief Title: Plastic Hat Trial to Prevent Hypothermia in Preterm Newborns in the Delivery Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Myra Wyckoff, Professor of Pediatrics, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 052008-049
Record Dates: First submitted 2009-02-27; First posted 2009-05-19 (Estimated); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Hypothermia
Keywords: hypothermia; euthermia; hyperthermia; mortality; morbidity; sepsis; bronchopulmonary dysplasia; intraventricular hemorrhage; ventilator days
MeSH Terms: conditions — Hypothermia; Hyperthermia; Sepsis; Bronchopulmonary Dysplasia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Plastic Cap (Experimental): Plastic lined stockinet cap (polyethylene bag)
  Interventions: Other: placement of plastic cap during delivery room stabilization
- Stockinet Cap (Active Comparator): Usual practice
  Interventions: Other: placement of routine cap during delivery room stabilization

INTERVENTIONS:
Other: placement of plastic cap during delivery room stabilization — placement of plastic cap during delivery room stabilization
  Arms: Plastic Cap
Other: placement of routine cap during delivery room stabilization
  Arms: Stockinet Cap

SUMMARY:
The purpose of this research project is to ascertain the effectiveness of plastic head covering in prevention of hypothermia. Hypothermia is defined by body temperature <36.5º Celsius by the World Health Organization. The surface area of the head is about 20% of total body surface of a newborn infant and is a major source of heat loss. The objective is to compare rectal temperature upon admission to the neonatal intensive care between preterm neonates who had stockinet head covering and those who had plastic-lined stockinet head covering placed in the delivery room. The investigators aim to demonstrate that plastic-lined head covering is more effective than stockinet head covering alone in maintaining body temperature.

DETAILED DESCRIPTION:
A prospective randomized control trial will be conducted in Parkland Memorial Hospital (PMH) neonatal intensive care unit (NICU) Dallas, Texas. Consent will not be obtained since: placement of plastic and/or stockinet head covering on the neonate is part of routine resuscitation care at PMH and by Neonatal Resuscitation Program (NRP) minimal risk to the preterm neonate is involved, post-delivery consent will be of little value since intervention only last ~24minutes, and obtaining informed consent from a mother who has labor pains or is on pain medication may be difficult.

Randomization of the neonates will be carried out in the delivery room by opening a sealed, opaque envelope just prior to birth. Qualified preterm newborns will be stratified into 2 OB EGA groups: (≤28weeks obstetrical(OB)estimated gestational age (EGA) and 29-32weeks OB EGA. In each stratified group, the newborns will be further randomized to control arm (stockinet head covering) or the intervention arm (plastic-lined head covering). Each arm of the study will have a sample size of 65, allowing for 130 infants in each OB EGA stratified group and for a sample size total of 260. Treatment versus control will be assigned by blocks of 8 by using a random permutation table. The assignment will be sealed in an opaque envelope by a non-participant person of the research.

The PMH high-risk resuscitation (RESUS) team attends all deliveries of infants ≤32 weeks OB EGA. The RESUS team is comprised of a resuscitation nurse, a respiratory therapist, and a practitioner. Neonatology fellow and/or attending may also attend these deliveries.

The use of warming aids by the RESUS team is standardized in the following manner: Randomization envelope will be opened. All infants will be taken from the obstetrician by the practitioner to an Ohio radiant warmer that has been pre-warmed to 100% capacity prior to the delivery of the infant. A food-grade storage (polyethylene) bag (will be referred as "poncho") will be used on all infants with the EGA of 32 weeks or less OB EGA to decrease evaporative and convective heat loss. The poncho will be placed by cutting a hole at the closed end of the bag for the purposes of inserting the head through it. The infants will not be dried except for the face as recommended by NRP. All infants that are ≤28weeks OB EGA will have a transwarmer mattress gel pad activated and placed on the radiant warmer during resuscitation and during transport as per PMH NICU and NRP standard practice. The appropriate head covering will then be placed to the level of the forehead on the infant as per randomization assignment. If access to the infant's umbilical cord is needed, a hole will be cut at the appropriate location. All infants will be transported in a dedicated isolette for resuscitation that has been prewarmed to 38ºC. The warming aids will be in place until the infant's arrival in the NICU.

The RESUS team will gather the following data in the delivery room: environmental temperature of the delivery room, rectal temperature immediately after delivery, annotation of warming aids implemented. The RESUS team also cares for the infant in the first 4 hours of life. Initial vital signs (heart rate, respiratory rate, and blood pressure), temperature, need of ventilation, need of intervention will be recorded by the RESUS team. After 4 hours the care will be assumed by the primary NICU team as per our standard practice.

Once the admission rectal temperature is taken, the head coverings will be removed and the infant will no longer be actively enrolled in the research. The rest of the data will be gathered through the Neonatal Resuscitation Database and Parkland NICU Morbidity and Mortality Database.

The rationale of this study is that no randomized control trial has been done to demonstrate the effectiveness of placement of plastic-lined head covering versus stockinet head covering. It would seem logical that if measures are taken to decrease heat loss from the head, these measures would improve temperature stability and avoid hypothermia in the premature neonate.

ELIGIBILITY:
Inclusion Criteria:

* Infants with less than 33 week gestational age by obstetrical dating
* Infants delivered in Parkland Memorial Hospital Labor and Delivery areas
* Infant whose delivery was attended by the Parkland Neonatal Resuscitation Team
* Infant whos is viable

Exclusion Criteria:

* Infant who has 33 week gestational age or greater by obstetrical dating
* Infant who is deemed non-viable
* Infant who did not have the Parkland Neonatal Resuscitation Team present at time of birth
* Infant with congenital anomaly which precludes measurement of rectal temperature (such as anal atresia or imperforate anus)

Max Age: 1 Hour | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 260 (Actual)
Dates: Start 2008-09 (Actual); Primary Completion 2010-09 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Hypothermia | 1 hour
  admission rectal temperature <36.5C

SECONDARY OUTCOMES:
Mortality | 1 year
  Death before hospital discharge
Infection | 1 year
  + blood cultures
Necrotizing enterocolitis | 1 year
  Bell Bell's criteria
Intraventricular Hemorrhage | 1 year
  Any grade
Bronchopulmonary Dysplasia | 1 year
  Oxygen requirement at 36 weeks corrected age (NIH definition)
Days on Ventilator | 1 year
  Invasive ventilation
Length of hospital stay | 1 year
  days of initial hospitalization after birth

CONTACTS AND LOCATIONS:
Overall Officials: Lilian T StJohn, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- Parkland Memorial Hospital, Dallas, Texas, United States